CLINICAL TRIAL: NCT01881724
Title: Impact of Sleep Education Program on Glycemic Control in Hong Kong Chinese Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Alice Pik Shan KONG, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUHK466711
Record Dates: First submitted 2011-10-18; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention)
- sleep education program (Experimental)
  Interventions: Behavioral: Sleep education

INTERVENTIONS:
Behavioral: Sleep education
  Arms: sleep education program

SUMMARY:
This is a randomized controlled trial with 12 month sleep education as intervention, followed by a 12 month observational period, to study whether sleep education would improve glycemic control and cardiometabolic profile of sleep deprived type 2 diabetic patients and evaluate the neurohormonal changes associated with sleep education.

DETAILED DESCRIPTION:
Patients will be identified from the Diabetes Mellitus and Endocrine Centre of Prince of Wales Hospital and Yao Chung Kit Diabetes Assessment Centre, The Chinese University of Hong Kong. All participants will have diabetes complications screening and comphrensive evaluations for glycemic control and cardiometabolic risk factors.Eligible subjects will be randomized to 2 groups (usual or conventional care versus intervention with sleep education program) for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Type 2 diabetes mellitus
3. Chinese ethnicity
4. Able and willing to give informed written consent
5. Sleep deprived, defined as subjective sleeping time <6 hours per day

Exclusion Criteria:

1. Type 1 diabetes mellitus
2. Known history of psychiatric disorders (e.g. depression, anxiety, dementia)
3. Sleep disorders secondary to another medical condition (e.g. obstructive sleep apnoea (OSA), circadian rhythm sleep disorder)
4. Concomitant chronic medical condition that was likely to be the cause of sleep problem (e.g. benign prostatic hypertrophy, chronic pain)
5. Concurrent use of hypnotic drugs, psychotic medications and any drugs that are known to affect sleep.
6. Any condition, as judged by the investigators, as ineligible to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from baseline | 12 months

SECONDARY OUTCOMES:
fasting plasma glucose | 12 months
insulin resistance | 12 months
  HOMA_IR
body weight | 12 months
blood pressure | 12 months
lipid profile | 12 months
sleep duration | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alice PS Kong, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- The Chinese University of Hong Kong, Hong Kong, China
- Clinical Trial Centre, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong